CLINICAL TRIAL: NCT00098254
Title: Phase II Study of Bay 43-9006 (Sorafenib) With Evaluation of RAS Signal Pathway in Patients With Relapsed Non-Small Cell Lung Cancer
Brief Title: BAY 43-9006 (Sorafenib) to Treat Relapsed Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Giuseppe Giaccone, M.D./National Cancer Institute, National Institutes of Health
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 050049; 05-C-0049; NCT00100763 (obsolete NCT alias)
Record Dates: First submitted 2004-12-03; First posted 2004-12-06 (Estimated); Results first posted 2012-05-02 (Estimated); Last update posted 2012-05-02 (Estimated); Status verified 2012-04

CONDITIONS: Non-Small-Cell Lung Carcinoma
Keywords: Non-Small Cell; Molecular; Targeted; Therapies; Cancer; Non-Small Cell Lung Cancer; NSCLC
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Neoplasms | interventions — Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- BAY 43-9006 (Sorafenib) (Experimental): Self administered oral doses at 400 mg twice a day with 250 ml (8 oz.) of water each morning and evening (i.e., 12-hourly) continuously in a 28 day cycle. Tablets may be taken with or without food.
  Interventions: Drug: BAY 43-9006 (Sorafenib)

INTERVENTIONS:
Drug: BAY 43-9006 (Sorafenib) — Self administered oral doses at 400 mg twice a day with 250 ml (8 oz.) of water each morning and evening (i.e., 12-hourly) continuously in a 28 day cycle. Tablets may be taken with or without food.
  Other Names: Sorafenib tosylate

SUMMARY:
This study will investigate the effects and side effects of BAY 43-9006 in patients with advanced, recurrent, or refractory non-small cell lung cancer (NSCLC). BAY 43-9006 is one of a new class of anticancer agents known as bi-aryl ureas.

Patients 18 years of age and older with NSCLC that has recurred or progressed after one regimen of chemotherapy may be eligible for this study. Candidates are screened with a medical history and physical examination; blood tests; tumor biopsy (see below); chest x-ray; electrocardiogram; and imaging studies, including positron emission tomography-computed tomography (PET-CT, see below) and dynamic, contrast-enhanced MRI (DCE-MRI, see below).

Participants take BAY 43-9006 by mouth twice a day, morning and evening. On the first and 15th days of treatment, patients are admitted to the hospital for pharmacokinetic studies; that is, a test of how the body handles the drug. For the test, blood is collected at intervals (at 15 minutes, 30 minutes, and 1, 2, 4, 6, 8, 12 and 24 hours after ingestion) to determine the drug's level in the bloodstream. Treatment with BAY 43-9006 continues until the study doctor determines that the medication is not beneficial or the patient wishes to withdraw from the study.

In addition to drug therapy, patients undergo the following tests and procedures:

* Physical examination every 4 weeks
* Blood pressure checks once a week during the first 4 weeks
* Blood tests every week
* CT scans or other imaging tests, such as ultrasound or MRI, every 8 weeks to evaluate the tumor's response to treatment. CT is an x-ray test that provides detailed pictures of the inside of the body. It can be done from different angles, providing a 3-dimensional picture of the part of the body being studied and allowing the doctor to see the location, nature, and extent of disease. MRI uses a powerful magnet and radio waves instead of x-rays to produce accurate, detailed pictures of organs and tissues.
* PET-CT approximately every 8 weeks to look at how different parts of the body take up and use glucose (a sugar nutrient). Because rapidly growing cells, such as tumors, use more sugar than normal cells do, this test can be used to detect cancer. For the test, the patient is given an injection of a sugar solution in which a radioactive tracer has been attached to the sugar molecule. A special camera detects the radiation emitted by the solution, and the resulting images show how much sugar is being used in various parts of the body. PET-CT uses the PET scan in combination with standard CT in a machine that does both tests.
* DCE-MRI after 2 weeks of treatment. This test uses MRI with a special non-radioactive dye to examine blood flow in a certain part of the body.
* Tumor biopsy (optional) after 2 weeks of treatment. A biopsy is the surgical removal of a small piece of tissue. The tumor biopsy is done either using a small bore needle under CT guidance or by direct visualization using a laparoscope/thoracoscope. For the needle biopsy, a needle is inserted through the skin and guided by CT into the tumor mass. For the laparoscopy/thoracoscopy, the patient is sedated or asleep and small lighted tubes are inserted into small holes made in the skin. The tumor is located and tissue withdrawn.

DETAILED DESCRIPTION:
Despite advances in systemic chemotherapy, patients with stage IV NSCLC will die from their disease. The median survival of all patients is 8-16 months, with a one year-survival rate of 33%. Chemotherapy is the mainstay of treatment of advanced disease. Based on available data from randomized trials, current treatment recommendations are to treat with one of several effective cisplatin-doublets which have resulted in median survival of 16 to 18 months. Second line chemotherapy is able to improve outcome in patients who have had prior cisplatin therapy. Although these important milestones represent improvements in the care of patients with metastatic NSCLC, outcome has not been able to be further improved by substituting one active drug for another in a platinum-based doublet, treating patients with more than four cycles of chemotherapy or by using cisplatin-based triplets. It is clear that if we are to improve outcome of NSCLC patients, we will need to develop drugs with novel mechanisms of action that perhaps will inhibit major cellular signaling pathways affecting survival, proliferation and angiogenesis. One new compound, BAY 43-9006, was designed to inhibit Raf and is also known to inhibit other kinases including VEGFR2, VEGFR3, PDGFR-beta, Flt3, c-KIT, and p38(1). BAY 43-9006 has shown in vitro activity against NSCLC cell lines NCI-H460 and A549 with tumor growth inhibition of 27% to 68%. In addition, BAY 43-9006 has shown activity in the H460 NSCLC xenograft model. In NSCLC, the proliferation signaling of the Ras/Raf/MEK/ERK pathway is increased due to the frequent (30%) presence of K-ras mutations in the tumor. Mutations in K-ras have been associated with malignant transformation of normal epithelium and constitutive activation of p21 and its downstream effects on cellular proliferation and inhibition of apoptosis. Clinical observations have shown that tumors with K-ras mutations tended to be smaller but more poorly differentiated, and associated with a significantly worse three-year mortality rate. As mentioned above, other pathways significant to the malignant potential of NSCLC, particularly those involved in angiogenesis, may also be affected by BAY 43-9006. The in vitro and in vivo data support the clinical investigation of BAY 43-9006 as an inhibitor of the Ras/Raf/MEK/ERK downstream proliferation effects. The goal of this phase II trial is to determinate if BAY 43-9006 is active in NSCLC, and to measure the BAY 43-9006 biological effects on the Ras/Raf/MEK/ERK pathway. To achieve these goals, patients with relapsed or recurrent NSCLC will be given BAY 43-9006 (four weeks cycle of 400mg PO BID). A series of correlative studies will be done during treatment to measure biological and clinical effects of BAY 43-9006. These studies will include analyses of tissue and blood samples as well as correlative imaging studies.

ELIGIBILITY:
* INCLUSION CRITERIA:

Histologically documented Non-small cell lung cancer and confirmed by the Laboratory of Pathology at the Clinical Center/National Institutes of Health (NIH) or the Laboratory of Pathology at National Naval Medical Center (NNMC).

Recurrent or progressed Non-Small Cell Lung Cancer (NSCLC).

Patients must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) as greater than 20 mm with conventional techniques or as greater than 10 mm with spiral Computed tomography (CT) scan.

Patients must have recovered from toxicity related to prior therapy to at least to grade 1 (defined by Common Terminology Criteria for Adverse Events (CTCAE) 3.0) and must not have had prior chemotherapy within 4 weeks. Patients must be at least 28 days since any prior radiation or major surgery.

Age greater than 18 years (males or non-pregnant females). Because no dosing or adverse event data are currently available on the use of BAY 43-9006 in patients less than 18 years of age, children are excluded from this study but will be eligible for future pediatric single-agent trials, if applicable.

Life expectancy of greater than 3 months.

Eastern Cooperative Oncology Group (ECOG) performance status less than 2 (Karnofsky > 60%).

Patients must have adequate organ and marrow function (as defined below). Patients must have returned to base line or grade one from any acute toxicity related to prior therapy.

Leukocytes greater than 3,000/micro l;

Absolute neutrophil count greater than 1,200/micro l;

Platelets greater than 100,000/micro l;

International normalized ratio (INR) less than or equal to 1.2

Partial thromboplastin time (PTT) less than or equal to 36 seconds or abnormality can be explained by the presences of lupus anticoagulant

Total bilirubin less than or equal to 1.5 times the institutional upper limits of normal;

Aspartate aminotransferase, oxaloacetic transaminase (AST,SGOT) and alanine transaminase, serum glutamic pyruvic transaminase (ALT,SGPT) less than 2.5 times the institutional upper limits of normal;

Creatinine or creatinine clearance less than or equal to 1.5 times the institutional upper limits of normal or greater than 45 mL/min/1.73 m^2 for patients with creatinine levels above institutional normal.

The effects of BAY 43-9006 on the developing human fetus at the recommended therapeutic dose are unknown. For this reason and because kinase inhibitors are known to be teratogenic, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation and continue for at least 2 months after completion. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with BAY 43-9006, breastfeeding should be discontinued if the mother is treated with BAY 43-9006.

Ability to comply with daily oral self administration schedule, and the ability to understand and the willingness to sign a written informed consent document.

EXCLUSION CRITERIA:

Patients with symptomatic brain metastases should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events. However, patients who have had treatment for their brain metastases and whose brain metastatic disease status has remained stable for at least 3 months without steroids may be enrolled at the discretion of the principal investigator.

Uncontrolled medical illness including, but not limited to, ongoing or uncontrolled, symptomatic congestive heart failure (American Heart Association (AHA) Class II or worse), uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.

Human immunodeficiency virus (HIV)positive patients receiving combination anti-retroviral therapy are excluded from the study because of possible pharmacokinetic interactions with BAY 43-9006. HIV positive patients not receiving antiretroviral therapy are excluded due to the possibility that BAY 43-9006 may worsen their condition and the likelihood that the underlying condition may obscure the attribution of adverse events with respect to BAY 43-9006.

Patients may not be receiving any other investigational agents.

History of another invasive malignancy in the last five years. Non-invasive, non-melanoma skin cancers will be allowed.

Patients with conditions that would impair their ability to swallow tablets are excluded.

Patients must not have any evidence of bleeding diathesis.

Patients must not be on therapeutic anticoagulation. Prophylactic anticoagulation (i.e. low dose warfarin) of venous or arterial access devices is allowed provided that the requirements for prothrombin time (PT), international normalized ratio (INR) or partial thromboplastin time (PTT) are met.

Both men and women and members of all races and ethnic groups are eligible for this trial. Every effort will be made to recruit women and minorities in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2004-12; Primary Completion 2009-11 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Giaccone, M.D., Ph.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Schiller JH, Harrington D, Belani CP, Langer C, Sandler A, Krook J, Zhu J, Johnson DH; Eastern Cooperative Oncology Group. Comparison of four chemotherapy regimens for advanced non-small-cell lung cancer. N Engl J Med. 2002 Jan 10;346(2):92-8. doi: 10.1056/NEJMoa011954. PMID 11784875
- [Background] Scagliotti GV, De Marinis F, Rinaldi M, Crino L, Gridelli C, Ricci S, Matano E, Boni C, Marangolo M, Failla G, Altavilla G, Adamo V, Ceribelli A, Clerici M, Di Costanzo F, Frontini L, Tonato M; Italian Lung Cancer Project. Phase III randomized trial comparing three platinum-based doublets in advanced non-small-cell lung cancer. J Clin Oncol. 2002 Nov 1;20(21):4285-91. doi: 10.1200/JCO.2002.02.068. PMID 12409326
- [Background] Choy H, Devore RF 3rd, Hande KR, Porter LL, Rosenblatt P, Yunus F, Schlabach L, Smith C, Shyr Y, Johnson DH. A phase II study of paclitaxel, carboplatin, and hyperfractionated radiation therapy for locally advanced inoperable non-small-cell lung cancer (a Vanderbilt Cancer Center Affiliate Network Study). Int J Radiat Oncol Biol Phys. 2000 Jul 1;47(4):931-7. doi: 10.1016/s0360-3016(00)00420-x. PMID 10863062
- [Result] Kelly RJ, Rajan A, Force J, Lopez-Chavez A, Keen C, Cao L, Yu Y, Choyke P, Turkbey B, Raffeld M, Xi L, Steinberg SM, Wright JJ, Kummar S, Gutierrez M, Giaccone G. Evaluation of KRAS mutations, angiogenic biomarkers, and DCE-MRI in patients with advanced non-small-cell lung cancer receiving sorafenib. Clin Cancer Res. 2011 Mar 1;17(5):1190-9. doi: 10.1158/1078-0432.CCR-10-2331. Epub 2011 Jan 11. PMID 21224376
- See also: NIH Clinical Center Detailed Web Page — http://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2005-C-0049.html
- See also: Medline Plus — http://www.nlm.nih.gov/medlineplus/
- See also: Drug Information — http://druginfo.nlm.nih.gov/drugportal/drugportal.jsp
- See also: US FDA Resources — http://www.clinicaltrials.gov/ct2/info/fdalinks
- See also: RECIST — http://ctep.cancer.gov/protocolDevelopment/docs/theasserecistjnci.pdf

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | BAY 43-9006 (Sorafenib)
Started | 37
Completed | 34
Not Completed | 3
Not completed — Adverse Event | 2
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Arm/Group | BAY 43-9006 (Sorafenib)
Number analyzed (Participants) | 37
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 20
  >=65 years | 17
Age Continuous [Mean (Standard Deviation); unit: years] | 61.9 (12.19)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 18
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 4
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 26
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 37

OUTCOME MEASURES:

1. Primary Outcome: Response Rate
Description: Percentage of participants with response rate = CR + PR. Response will be evaluated by the Response Evaluation Criteria in Solid Tumors (RECIST) criteria. CR (complete response) is the disappearance of all target lesions; PR (partial response) is a 30% decrease in the sum of the longest diameter of target lesions; PD (progressive disease) is a 20% increase in the sum of the longest diameter of target lesions; and SD (stable disease) are small changes that do not meet the above criteria. Please see the Protocol Link module for additional information about RECIST if desired.
Time Frame: 17 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | BAY 43-9006 (Sorafenib)
Number analyzed (Participants) | 34
percentage of participants | 6 [1 to 20]

2. Primary Outcome: Progression Free Survival
Description: Time between the first day of treatment to the day of disease progression. Progressive disease is at least a 20% increase in the sum of the longest diameter of target lesions.
  Appearance of one or more new lesions and/or unequivocal progressions of existing non-target lesions.
Time Frame: 17 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | BAY 43-9006 (Sorafenib)
Number analyzed (Participants) | 34
months | 3.4 [1.9 to 3.7]

3. Primary Outcome: The Number of Participants With Adverse Events
Description: Here are the total number of participants with adverse events. For the detailed list of adverse events see the adverse event module.
Time Frame: 5 1/2 years
Measure: Number; unit: Participants
Arm/Group | BAY 43-9006 (Sorafenib)
Number analyzed (Participants) | 37
Participants | 37

4. Secondary Outcome: Overall Survival
Description: Time between the first day of treatment to the days of death.
Time Frame: 17 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | BAY 43-9006 (Sorafenib)
Number analyzed (Participants) | 34
months | 11.6 [9.2 to 16.4]

5. Secondary Outcome: Percent of Participants With Genotyping of CYP3A4/5 and 5 Polymorphisms
Description: All patients will be genotyped for CYP3A4/5 and 5 polymorphisms.
Time Frame: 58 months
Population: The analysis for this outcome measure was not performed. Endpoint lost interest when mutation analysis was felt to be more important.
Measure: Number; unit: Percent of participants
Arm/Group | BAY 43-9006 (Sorafenib)
Number analyzed (Participants) | 0

6. Secondary Outcome: Overall Survival Reported Separately for Participants With a Change in PLGF Below 11 pg/ml and Above 12 pg/ml
Description: Difference in placental derived growth factor (PLGF) between day 28 and day 0 of < 11 pg/ml vs. > 12 pg/ml.
Time Frame: 17 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | BAY 43-9006 (Sorafenib)
Number analyzed (Participants) | 37
months
  PLGF ,< 11 pg/ml | 6.6 [4.9 to 9.2]
  PLGF > 12 pg/ml | 15.6 [9.4 to 22.5]
Statistical Analysis 1: Comparison: BAY 43-9006 (Sorafenib); Test type: Superiority or Other; p = 0.0027, Kaplan-Meier

7. Secondary Outcome: Cytokine Levels
Description: Serial plasma samples were collected from all patients and cytokine levels were measured. The concentrations of the cytokines were determined with recombinant standards and expressed as picograms per milliliter (pg/ml).
Time Frame: 54 days
Measure: Median (Inter-Quartile Range); unit: pg/ml
Arm/Group | BAY 43-9006 (Sorafenib)
Number analyzed (Participants) | 37
pg/ml
  VEGF | 101 [69 to 204]
  sVEGFRI | 115 [91 to 198]
  PLGF | 19 [12 to 29]
  bFGF | 6 [2.9 to 14]

8. Secondary Outcome: Correlation of Response to Treatment With KRAS Mutational Status
Description: Mutational analysis of these genes was performed on paraffin-imbedded tissue blocks from prior pathologic specimens. Disease control rate was correlated with KRAS mutational status. Disease control rate was defined as complete remission (CR) + partial remission (PR)+ stable disease (SD).
Time Frame: 42 months
Population: 11/34 KRAS positive; 23/34 KRAS negative 5/23 EGFR positive; 18/23 EGFR negative
Measure: Number; unit: percentage of participants
Arm/Group | BAY 43-9006 (Sorafenib)
Number analyzed (Participants) | 37
percentage of participants
  DCR observed in KRAS mutant participants | 60
  DCR observed in KRAS wild-type participants | 71
  DCR observed in EGFR mutant participants | 40
  DCR observed in EGFR wild-type participants | 69
Statistical Analysis 1: Comparison: BAY 43-9006 (Sorafenib); Test type: Superiority or Other; p = 0.33, Kaplan-Meier

9. Secondary Outcome: Overall Survival Associated With Basic Fibroblast Growth Factor (bFGF)
Description: Serum plasma is collected at the beginning of each cycle during the course of the study and analyzed by the enzyme-linked immunosorbent assay (ELISA).
Time Frame: 42 months
Population: 14 patients with day 28 FGF >6 and 14 patients with FGF <6.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | BAY 43-9006 (Sorafenib)
Number analyzed (Participants) | 14
months
  Overall survival for bFGF day 0<6 pg/ml | 15.4 [9.2 to 31.2]
  Overall survival for bFGF day 0>6 pg/ml | 5.5 [3.1 to 16.4]
Statistical Analysis 1: Comparison: BAY 43-9006 (Sorafenib); Test type: Superiority or Other; p = 0.042, Kaplan-Meier

10. Secondary Outcome: Progression Free Survival Associated With Basic Fibroblast Growth Factor (bFGF)
Description: as for outcome 9
Time Frame: 17 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | BAY 43-9006 (Sorafenib)
Number analyzed (Participants) | 14
months
  Progression free survival for bFGF day 28<6 pg/ml | 4.4 [3.1 to 5.5]
  Progression free survival for bFGF day 28>6 pg/ml | 1.8 [1.4 to 3.7]
Statistical Analysis 1: Comparison: BAY 43-9006 (Sorafenib); Test type: Superiority or Other; p = 0.028, Kaplan-Meier

11. Secondary Outcome: Percentage of Participants With an Increase or Decrease in the Reverse Contrast Transfer Rate (Kep), Forward Contrast Transfer Rate (Ktrans), and Extravascular Fraction (Ve) With the Dynamic Contrast Enhanced Magnetic Resonance Imaging (DCE-MRI)
Description: DCE-MRI was used to evaluate changes (e.g. decrease/increase in Ve, Ktrans, Kep value) in vascularity and quality of index lesions to provide early indication of treatment effect before changes in size can be perceived on CT. Changes were reflected in a decrease/increase of Ve, Ktrans, or Kep (Kep, Ve, Ktrans measurements at day 0, day 14 and the difference between the day 14 and the day 0 measurements (day 14-day 0).
Time Frame: 59 months
Measure: Number; unit: Percentage of participants
Arm/Group | BAY 43-9006 (Sorafenib)
Number analyzed (Participants) | 37
Percentage of participants
  percentage of pts with an increase in Ktrans orKep | 19
  percentage of pts with an decrease in Ktrans orKep | 81
  Percentage of pts with an increase or decrease-Ve | 0

12. Secondary Outcome: Percent of Participants Who Had Immunohistochemical Analysis Performed for Raf, MEK, ERK, ERK-1 and p90RSK,ERK, E Twenty-six (ETS)-Like Transcription Factor 1 (ELK-1) and p90Ribosomal S6 Kinase (p90RSK).
Description: Immunohistochemical analysis performed by using state specific antibodies against Raf, methyl ethyl ketone (MEK), extracellular-signal regulated kinase (ERK), and two downstream substrates of ERK, E twenty-six (ETS)-like transcription factor 1 (ELK-1) and p90Ribosomal S6 kinase (p90RSK).
Time Frame: 59 months
Population: The analysis for this outcome measure was not performed. Endpoint lost interest when mutation analysis was felt to br more important.
Measure: Number; unit: Percent of participants
Arm/Group | BAY 43-9006 (Sorafenib)
Number analyzed (Participants) | 0

13. Secondary Outcome: Percent of Participants Who Had Cytokine Profiling for IL-6 and IL-8
Description: Serial plasma samples were collected from all patients at pretreatment (baseline - day 0), and on days 14, 28, and 54. The concentrations of the cytokines were determined with recombinant standards and expressed as picograms per milliliter (pg/ml).
Time Frame: 60 months
Population: as for outcome 5
Measure: Number; unit: Percent of participants
Arm/Group | BAY 43-9006 (Sorafenib)
Number analyzed (Participants) | 0

14. Secondary Outcome: Percentage of Participants With BRAF Mutations
Description: Extracted DNA was subjected to an initial PCR using a single primer set encompassing codom V600. Pyrosequencing was carried out on a Qiagen PyroMaark Q24 system.
Time Frame: 60 months
Population: as for outcome 5
Measure: Number; unit: Percent of participants
Arm/Group | BAY 43-9006 (Sorafenib)
Number analyzed (Participants) | 0

15. Secondary Outcome: Percent of Pts With Primary Pharmacoproteomic Modulation Targets
Description: Pharmacoproteomic modulation targets (AKT, p-AKT, ERK 1/2, MEK, Cyclin D, p-ERK 1/2, p-MEK, pMEK, eNOA, p-eNOA, Cleaved PARP, PDGFRbeta, p-PDGFRbeta,Cyclin D, CD31, PARP. Caspase 9, Caspase 3, Cleaved Caspase-9 Cleaved Caspase 3)
Time Frame: 60 months
Population: as for outcome 5
Measure: Number; unit: mg/ml
Arm/Group | BAY 43-9006 (Sorafenib)
Number analyzed (Participants) | 0

16. Secondary Outcome: Secondary Pharmacoproteomic Modulation Targets
Description: Secondary pharmacoproteomic modulation targets (mTOR, EGFR, Src, NFkB, STAT1, TGFa, p38, Jak 1, lkB, IGFR, p-mTOR, p-EGFR, p-Src, p-NFkB, p-STAT1, Phospho-p38, p-Jak1, p-lkB,Pyk2, p-Pyk2, VEGFR-2, GSK3beta, p-GSK3beta, p-bad, p-Bcl-2, PCNA, Fos, Raf, CREB, Rho, avbeta3complex, Bad, CD34, VEGFR-1, bfGF, vWF, Factor VIII, Annexin V, Bcl-2).
Time Frame: 60 months
Population: as for outcome 5
Measure: Number; unit: mg/ml
Arm/Group | BAY 43-9006 (Sorafenib)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 5 years, 6 months, and 21 days
Arm/Group | BAY 43-9006 (Sorafenib)
Serious Adverse Events (participants affected / at risk) | 11/37
Other Adverse Events (participants affected / at risk) | 37/37
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BAY 43-9006 (Sorafenib) (N=37)
Alanine aminotransferase increased (Investigations) | 1 (2)
Alkaline phosphatase increased (Investigations) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 1 (4)
Aspartate aminotransferase increased (Investigations) | 1 (2)
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Confusion (Psychiatric disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Death NOS (General disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4 (5)
Fatigue (General disorders) | 1 (1)
Hypermagnesemia (Metabolism and nutrition disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (2)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (3)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (2)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Lung infection (Infections and infestations) | 2 (4)
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 (3)
Platelet count decreased (Investigations) | 1 (4)
Vasculitis (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BAY 43-9006 (Sorafenib) (N=37)
Activated partial thromboplasstin time prolonged (Investigations) | 14 (20)
Alanine aminotransferase increased (Investigations) | 12 (17)
Alkaline phosphatase increased (Investigations) | 9 (12)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 3 (3)
Creatinine increased (Investigations) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 13 (23)
Anorexia (Metabolism and nutrition disorders) | 9 (12)
Anxiety (Psychiatric disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 18 (42)
Ataxia (Nervous system disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (4)
Blood bilirubin increased (Investigations) | 7 (11)
Blood prolactin abnormal (Investigations) | 1 (1)
Blurred vision (Eye disorders) | 3 (3)
Bronchopulomonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 2 (2)
CPK increased (Investigations) | 4 (7)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Chills (General disorders) | 3 (3)
Confusion (Psychiatric disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 3 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 10 (14)
Dehydration (Metabolism and nutrition disorders) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 15 (29)
Dizziness (Nervous system disorders) | 4 (4)
Dry skin (Skin and subcutaneous tissue disorders) | 7 (7)
Dysgeusia (Nervous system disorders) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 2 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 6 (9)
Edema limbs (General disorders) | 2 (2)
Enterocolitis infections (Infections and infestations) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Fatigue (General disorders) | 11 (13)
Fever (General disorders) | 2 (3)
Flashing lights (Eye disorders) | 1 (1)
Flushing (Vascular disorders) | 2 (2)
Headache (Nervous system disorders) | 5 (8)
Hemoglobinuria (Renal and urinary disorders) | 1 (1)
Hot flashes (Vascular disorders) | 1 (1)
Hypercalcemia (Metabolism and nutrition disorders) | 6 (7)
Hyperglycemia (Metabolism and nutrition disorders) | 10 (22)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1)
Hyperkalemia (Metabolism and nutrition disorders) | 12 (22)
Hypermagnesemia (Metabolism and nutrition disorders) | 12 (17)
Hypernatremia (Metabolism and nutrition disorders) | 1 (2)
Hypertension (Vascular disorders) | 15 (20)
Hyperuricemia (Metabolism and nutrition disorders) | 2 (4)
Hypoalbuminemia (Metabolism and nutrition disorders) | 20 (35)
Hypocalcemia (Metabolism and nutrition disorders) | 4 (12)
Hypoglycemia (Metabolism and nutrition disorders) | 3 (3)
Hypokalemia (Metabolism and nutrition disorders) | 5 (7)
Hypomagnesemia (Metabolism and nutrition disorders) | 10 (15)
Hyponatremia (Metabolism and nutrition disorders) | 17 (41)
Hypophosphatemia (Metabolism and nutrition disorders) | 20 (44)
Hypotension (Vascular disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
INR increased (Investigations) | 1 (1)
Insomnia (Psychiatric disorders) | 3 (3)
Investigations-Other, specify (Investigations) | 1 (1) — Bicarbonate, serum-low
Lipase increased (Investigations) | 3 (4)
Lung infection (Infections and infestations) | 1 (1) — Pulmonary infiltrates
Lung infection (Infections and infestations) | 3 (3)
Lymphocyte count decreased (Investigations) | 16 (37)
Mucositis oral (Gastrointestinal disorders) | 7 (13)
Myalgia (Musculoskeletal and connective tissue disorders) | 5 (6)
Nausea (Gastrointestinal disorders) | 8 (13)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Nervous system disorders-Other, specify (Nervous system disorders) | 1 (1) — JITTERS
Neutrophil count decreased (Investigations) | 3 (10)
Non-cardiac chest pain (General disorders) | 2 (3)
Otitis externa (Ear and labyrinth disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 (5)
Palmar-plantar erythrodyesthesia syndrome (Skin and subcutaneous tissue disorders) | 23 (69)
Pericardial effusion (Cardiac disorders) | 1 (1)
Peripheral motor neuropathy (Nervous system disorders) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 5 (5)
Pharyngitis (Infections and infestations) | 1 (1)
Platelet count decreased (Investigations) | 11 (15)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pruritis (Skin and subcutaneous tissue disorders) | 7 (8)
Rash maculopaular (Skin and subcutaneous tissue disorders) | 20 (30)
Respiratory, thoracic and mediastinal disorders-Other, specify (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Cold
Retinopathy (Eye disorders) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 2 (2)
Sinusitis (Infections and infestations) | 1 (1)
Skin and subcutaneous tissue disorders-Other, specify (Skin and subcutaneous tissue disorders) | 1 (1) — Warts Lt forearm
Skin and subcutaneous tissue disorders-Other, specify (Skin and subcutaneous tissue disorders) | 1 (1) — keratocanthoma
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 (1)
Thromboembolic event (Vascular disorders) | 1 (1)
Treatment related secondary malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Tremor (Nervous system disorders) | 1 (1)
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Urinary frequency (Renal and urinary disorders) | 1 (1)
Uterine hemorrhage (Reproductive system and breast disorders) | 1 (1)
Vaginal infection (Infections and infestations) | 1 (1)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 1 (4)
Skin and subcutaneous tissue disorders-Other, specify (Skin and subcutaneous tissue disorders) | 1 (1) — Possible keratoacanthoma
Syncope (Nervous system disorders) | 1 (1)
Serum amylase increased (Investigations) | 3 (6)
Vomiting (Gastrointestinal disorders) | 3 (6)
Weight loss (Investigations) | 5 (9)
White blood cell decreased (Investigations) | 7 (15)
Wound dehiscence (Injury, poisoning and procedural complications) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No